CLINICAL TRIAL: NCT01179932
Title: Acute Anesthesia Charting Fidelity Quality Assessment Pilot Study
Brief Title: Anesthesia Charting Fidelity Study
Status: Withdrawn | Type: Observational
Why Stopped: Never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Edwin Avery, Principle Investigator, University Hospitals
Other Study IDs: Charting Pilot
Record Dates: First submitted 2010-07-26; First posted 2010-08-11 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia
Keywords: Pilot; Charting; Anesthesia Record; Cardiac surgical operating room; Cardiac surgical intensive care unit; Electrophysiology lab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anesthesia Record: The nursing and anesthesia records will be examined for accuracy and completeness
  Interventions: Other: No Intervention Used

INTERVENTIONS:
Other: No Intervention Used — Our study is observational; therefore, there is no type of intervention being used.

SUMMARY:
Primary Objective: Conduct a prospective, observational pilot study that assesses the frequency and severity of anesthesia charting fidelity weaknesses in three separate clinical environments (Cardiac surgical operating room, cardiac surgical intensive care unit, and electrophysiology laboratory) as assessed by a customized error scoring system that focuses on the magnitude of errors among multiple continuous, categorical and dichotomous variables. The errors are being assessed in order to identify the most common charting inaccuracies so that target areas appropriate for testing of improvement strategies may be isolated.

DETAILED DESCRIPTION:
1. Primary Objective: Conduct a prospective, observational pilot study that assesses the frequency and severity of anesthesia charting fidelity weaknesses in three separate clinical environments (Cardiac surgical operating room, cardiac surgical intensive care unit, and electrophysiology laboratory) as assessed by a customized error scoring system that focuses on the magnitude of errors among multiple continuous, categorical and dichotomous variables. The errors are being assessed in order to identify the most common charting inaccuracies so that target areas appropriate for testing of improvement strategies may be isolated.

   1. Cardiac surgical operating room: Any cardiac surgical procedure that involves the use of cardiopulmonary bypass and planned postoperative intensive care unit admission in an electronic supplemented anesthesia charting environment
   2. Cardiac surgical intensive care unit: The cardiac surgical intensive care unit environment during the first 2-3 hours following procedures referenced in section I,A,1
   3. Electrophysiology laboratory: select electrophysiology laboratory based procedures that employ a paper anesthesia chart
2. Secondary and Exploratory Objectives:

   1. Identify environmental variables that contribute significantly to medical record errors.
   2. Identify clinical role of individual responsible for charting
   3. Investigate time of day/patterns that charting errors occur
   4. Relationship of clinical acuity and event occurrences
   5. Role of equipment malfunction and event frequency
   6. Role of social distracters and event frequency
   7. Role of monitor infidelity and event frequency
   8. Role of delayed charting of event and frequency of errors
   9. Identify/quantify the awareness of clinicians to their execution of medical record errors through use of simple, multiple choice 4 question survey that clinicians will be asked to fill out following a case study
   10. Examine the relationship between the assessed environments and the frequency of medical charting errors
   11. Identify the areas of anesthesia charting most in need of improvement in order to address designing ways to potentially improve these weaknesses.

Error scoring system:

1. The degree of charting fidelity error in this study will be converted via a classification system to make data analysis more efficient. All types of errors that involve continuous variables will be assessed with mean, median and standard deviation as well as range. Numerical data points related to time will be classified into four separate categories.

   1. Class It: temporally accurate data will less than 2 minutes or 3.3% deviation from actual time of event/observation.
   2. Class IIt: temporally inaccurate data with between 2-3 minutes or 3.3-5% deviation from actual time of event/observation.
   3. Class IIIt: temporally inaccurate data with between 3-6 minutes or 5-10% deviation from actual time of event/observation.
   4. Class IVt: temporally inaccurate data with greater than 10% deviation (6 min) from actual time of event/observation.
2. The degree of charting fidelity error observed with respect to hemodynamic parameters will be classified as follows:

   1. Class Ih: accurate hemodynamic data with less than 3% deviation from the representative value recorded by the scribe.
   2. Class IIh: inaccurate hemodynamic data with between 3-5% deviation from the representative value recorded by the scribe.
   3. Class IIIh: inaccurate hemodynamic data with between 5-10% deviation from the representative value recorded by the scribe.
   4. Class IVh: inaccurate hemodynamic data with greater than 10% deviation from the representative value recorded by the scribe.
3. The degree of charting fidelity error observed with respect to whether a procedure which was performed by anesthesia provider was charted will be assessed as a dichotomous variable, Yes or No.
4. The degree of charting fidelity error observed with respect to whether a significant intraoperative event, or intra-procedural event for the electrophysiology laboratory, was charted will be assessed as a dichotomous variable, Yes or No.
5. The degree of charting fidelity error observed with respect to drug dosing will be assessed as a dichotomous variable, Yes or No.
6. The degree of charting fidelity error as related to procedural details will be assessed as a dichotomous variable, Yes or No.
7. Full statistical analysis making all possible comparisons of collected data will be performed with the assistance of a trained statistician.

ELIGIBILITY:
a. Inclusion criteria:

1. Male or female patients ≥ 18 years of age
2. Patients and the hospital staff that are caring for them, scheduled to undergo any cardiac surgical procedure that involves the use of both general anesthesia (with planned computer assisted charting using the PISCES system) and cardiopulmonary bypass, including postoperative intensive care unit monitoring -or- Patients and the hospital staff caring for them scheduled to undergo select electrophysiologic procedures (detailed below 1 - 3) involving the administration of general anesthesia in the electrophysiology laboratory with planned manual paper charting

   1. Defibrillation threshold testing using non-invasive programmed stimulation of an implantable cardiovertor defibrillator (ICD)
   2. Transesophageal echocardiography guided electrical cardioversion of patients with supraventricular arrhythmias
   3. Electrical cardioversion of patients with supraventricular arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Deidentified patients undergoing a cardiac surgical procedure or undergoing select electrophysiologic procedures as well as the corresponding clinical staff caring for them.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2010-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Frequency/severity of anesthesia charting fidelity weaknesses in cardiac care based clinical environments as assessed by an error scoring system. | A total of thirty separate anesthesia records will be inidividually assessed and compared to the data prospectively collected during each corresponding anesthetic (lasting an average of 5 hours in the OR and 45 min in the EP lab.
  A single dedicated observer with focused clinical education will continually scribe observations made with close attention to detail (e.g., time of event, drug administered, dose of drug, route of administration of drug) using a prospectively designed data collection tool. This record of events will then be compared to the clinician charted anesthesia record in order to assess the frequency and severity of errors ocurring within the anesthesia record. A customized scoring system will be employed to grade the observed errors noted in the anesthesia record.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin G Avery, MD, Principal Investigator — UH Case Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Chamisa I, Zulu BM. Setting the records straight--a prospective audit of the quality of case notes in a surgical department. S Afr J Surg. 2007 Aug;45(3):92, 94-5. PMID 17892187
- [Result] Ho MY, Anderson AR, Nijjar A, Thomas C, Goenka A, Hossain J, Curley PJ. Use of the CRABEL Score for improving surgical case-note quality. Ann R Coll Surg Engl. 2005 Nov;87(6):454-7. doi: 10.1308/003588405X60687. PMID 16263017
- [Result] Devitt JH, Rapanos T, Kurrek M, Cohen MM, Shaw M. The anesthetic record: accuracy and completeness. Can J Anaesth. 1999 Feb;46(2):122-8. doi: 10.1007/BF03012545. PMID 10083991
- [Result] Byrne AJ, Sellen AJ, Jones JG. Errors on anaesthetic record charts as a measure of anaesthetic performance during simulated critical incidents. Br J Anaesth. 1998 Jan;80(1):58-62. doi: 10.1093/bja/80.1.58. PMID 9505779
- [Result] Byrne AJ, Jones JG. Inaccurate reporting of simulated critical anaesthetic incidents. Br J Anaesth. 1997 Jun;78(6):637-41. doi: 10.1093/bja/78.6.637. PMID 9215012